CLINICAL TRIAL: NCT02680314
Title: Is More Than One Dose of Misoprostol Needed to Expedite Vaginal Delivery in a Patient With an Unripe Cervix?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Peter S. Bernstein, Prof., Maternal Fetal Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5341
Record Dates: First submitted 2016-01-22; First posted 2016-02-11 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn
Keywords: unripe cervix
MeSH Terms: interventions — Misoprostol; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Dose (Active Comparator): single dose of misoprostol
  Interventions: Drug: Misoprostol
- Multiple Dose (Active Comparator): multiple doses of misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Misoprostol, a prostaglandin, binds to myometrial cells to cause strong myometrial contractions leading to expulsion of tissue. This agent also causes cervical ripening with softening and dilation of the cervix.
  Other Names: cytotec, methotrexate

SUMMARY:
The goal of this study is to determine whether inducing labor with just one dose of misoprostol, followed by treatment with oxytocin, will still be effective enough to increase the chances of having a successful vaginal delivery as compared to using more than one dose of misoprostol, followed by treatment with oxytocin.

DETAILED DESCRIPTION:
This study involves a comparison of two different regimens of prostaglandin use for "cervical ripening" prior to induction of labor. Women admitted to the hospital for induction of labor who are found to have "unripe" cervixes at the time of admission, and who agree to participate in the study will be randomly assigned to one of two treatment groups. In one group, a single dose of 25 µcg of misoprostol will be administered vaginally and four hours later oxytocin induction will be started if clinically indicated. In the second group of women, repeat doses of misoprostol will be given every four hours up to six doses unless labor or cervical ripening occurs sooner. At this point, oxytocin will be started as needed. Success of vaginal delivery by 24 hours, time from initiation of protocol to delivery and cesarean section rates will be compared. Complications such as postpartum hemorrhage, episodes of tachysystole with fetal compromise and chorioamnionitis and endometritis will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman undergoing induction of labor
* Live singleton pregnancy ≥ 37 week gestation
* Bishop score < 6
* Category I fetal heart rate

Exclusion Criteria:

* Contraindications to vaginal delivery (e.g. vasa previa, placenta prevue,non-vertex presentation, umbilical cord prolapse, and active genital herpes infection.)
* Pregnancies complicated by major fetal anomalies
* Any contraindication to the use of misoprostol, including
* History of previous c-section or major uterine surgery
* Prior allergic reaction
* Category II or III fetal heart rate
* Regular uterine contractions ≥ 3 in a 10-minute period persistent for at least 30 minutes
* Estimated fetal weight < 10 percentile
* Premature rupture of membranes
* Age < 18 years old
* Women who do not have the capacity to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05-17 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Tropper, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Dose | Multiple Dose
Started | 120 | 123
Completed | 120 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose | Multiple Dose | Total
Number analyzed (Participants) | 120 | 123 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 123 | 243
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 123 | 243
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African | 38 | 44 | 82
  Hispanic | 57 | 53 | 110
  other | 25 | 26 | 51
Region of Enrollment [Number; unit: participants]
  United States | 120 | 123 | 243

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaginal Delivery Within 24 Hours
Description: To compare the rate of vaginal delivery within 24 hours in patients who receive a single dose of misoprostol versus those receiving multiple doses of this medication.
Time Frame: within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose | Multiple Dose
Number analyzed (Participants) | 120 | 123
Participants | 50 | 55

2. Secondary Outcome: To Determine the Interval From Initiation of Misoprostol to Delivery in Each Group
Description: To determine the interval from initiation of misoprostol to delivery in each group
Time Frame: within 24 hours from the initial intervention
Population: Minutes from initiation of misoprostol to delivery
Measure: Median (Inter-Quartile Range); unit: Median number of Minutes
Arm/Group | Single Dose | Multiple Dose
Number analyzed (Participants) | 120 | 123
Median number of Minutes | 1187 [695 to 1628] | 1321 [900.5 to 1735]
Statistical Analysis 1: Comparison: Single Dose vs Multiple Dose; Test type: Superiority; p = 0.202, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Single Dose | Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/123
Other Adverse Events (participants affected / at risk) | 0/120 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02680314/Prot_SAP_000.pdf